CLINICAL TRIAL: NCT05652543
Title: Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant SARS-CoV-2 Alpha/Beta/Delta/Omicron Variants S Trimer Protein Vaccine (SCTV01E) in a Vaccinated Population
Brief Title: A PhaseⅡ Study to Evaluate the Safety & Immunogenicity of SARS-CoV-2 Alpha/Beta/Delta/Omicron Variants COVID-19 Vaccine
Acronym: SCTV01E
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SCTV01E-01-CHN-1
Record Dates: First submitted 2022-12-12; First posted 2022-12-15 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: COVID-19 Pandemic
Keywords: COVID-19 Pandemic, Vaccine
MeSH Terms: conditions — COVID-19 | interventions — SCTV01C vaccine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Participants ≥3 years old who has received the recommended dose and immunization procedure of domestically approved COVID-19 vaccine, Participants in each group (including the first 15 participants in Group A and sentry participants in groups B and C) will be randomly inoculated with either SCTV01E or placebo (normal saline) according to 4:1, i.e. 200 participants in each group will receive SCTV01E and 50 participants will receive placebo (normal saline).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine group (Experimental): Participants ≥3 years old who have received the recommended dose and immunization procedure of domestically approved COVID-19 vaccine will receive vaccine (SCTV01E).
  Interventions: Biological: SCTV01E
- Placebo group (Placebo Comparator): Participants ≥3 years old who have received the recommended dose and immunization procedure of domestically approved COVID-19 vaccine will receive placebo (normal saline)
  Interventions: Biological: Placebo (normal saline)

INTERVENTIONS:
Biological: SCTV01E — Participants will be vaccinated with SCTV01E on Day 0, and safety and immunogenicity will be monitored for 180 days after vaccination.
  Arms: Vaccine group
Biological: Placebo (normal saline) — Participants will be vaccinated with Placebo (normal saline) on Day 0, and safety and immunogenicity will be monitored for 180 days after vaccination.
  Arms: Placebo group

SUMMARY:
This study is a randomized, double-blind, placebo-controlled Phase II clinical trial to evaluate the safety and immunogenicity of SCTV01E in population of different ages who have been vaccinated against COVID-19. A total of 750 participants ≥3 years old who have received the recommended dose and immunization procedure of domestically approved COVID-19 vaccines will be enrolled, including 250 participants ≥18 years old (group A), 250 participants aged 12-17 years old (group B), and 250 participants aged 3-11 years old (group C). The study will be carried out gradually according to the age of the participants from older to younger. Considering that SCTV01E in this study is the first clinical study in participants under 18 years old, 15 sentinel participants will be assigned to group B and 30 sentinel participants will be assigned to group C (including 15 aged 6-11 years old and 15 aged 3-5 years old).

The Primary end points are 1. The incidence and severity of solicited adverse events on days 0-7 after inoculation with SCTV01E. 2. IgG total antibody concentrations (ELISA) against SARS-CoV-2 prototype strains and neutralizing antibodies titer (Live virus neutraliztion antibody test) against SARS-CoV-2 Omicron variant at 28 days post-vaccination.

DETAILED DESCRIPTION:
Firstly, 250 participants will be randomly enrolled in group A, among which the first 15 participants will be observed for 7 days after receiving the study vaccine and assessed for safety by the DSMB. If the 15 participants do not meet the study suspension/termination criteria, 15 sentinel participants in group B will be enrolled. The sentinel participants in Group B will be observed for 7 days after receiving the study vaccine, and safety is assessed by the DSMB. If the sentinel participants in group B do not meet the study suspension/termination criteria, non-sentinel participants in Group B and 15 sentinel participants in Group C aged 6-11 years old will be enrolled at the same time. The 15 sentinel participants aged 6-11 years in group C will be observed for 7 days after receiving the study vaccine and assessed for safety by the DSMB. If the study suspension/termination criteria are not met, non-sentinel participants aged 6-11 years old in group C and 15 sentinel participants aged 3-5 years old in group C will be enrolled, and sentinel participants aged 3-5 years old in group C will be observed for 7 days after receiving the study vaccine. Safety will be assessed by the DSMB and non-sentinel participants aged 3-5 years old in Group C will be enrolled if study suspension/termination criteria are not met in sentinel participants aged 3-5 years old.

Participants in each group (including the first 15 participants in Group A and sentinel participants in groups B and C) will be randomly inoculated with either SCTV01E or placebo (normal saline) at a ratio of 4:1, i.e. 200 participants in each group will receive SCTV01E and 50 participants will receive placebo (normal saline).

Randomized stratification factors for group A are age (18-59 years vs. ≥60 years), past COVID-19 vaccination status (completion of baseline immunization vs. Completion of booster immunization), the last type of COVID-19 vaccine received (inactivated vs. other vaccines), and the duration of prior Informed consent form (ICF) signing (6-12 months vs. 12-24 months); Randomized stratification factor for group B are past COVID-19 vaccination (completion of baseline immunization vs. Completion of booster immunization), type of COVID-19 vaccine last received (inactivated vs. other vaccines) and time since ICF last received (6-12 months vs. 12-24 months); Random stratification factors for group C are age (3-5 years vs. 6-11 years), past COVID-19 vaccination (completion of baseline immunization vs. Completion of enhanced immunization), the last type of COVID-19 vaccine received (inactivated vs. other vaccines), and the duration of prior Informed consent form (ICF) signing (6-12 months vs. 12-24 months).

ELIGIBILITY:
Inclusion Criteria:

* The age when signing ICF should meet the requirements of the scheme (Group A ≥18 years old; Group B 12-17 years old; Group C, 3-11 years old) male or female;
* Have previously received the recommended dose and immunization procedures of COVID-19 vaccine approved for domestic market, and the interval between signing ICF and receiving the last dose of COVID-19 vaccine is 6-24 months;
* Subject and/or guardian or client of both parties are able to sign a written ICF and voluntarily participate in the trial, fully understand the trial procedure, the risks of participating in the trial and the alternative interventions available to non-participants;
* The subject and/or the guardian or client of both parties can read, understand and fill in the diary card;
* Healthy subjects or subjects with stable underlying diseases. Stable underlying diseases were defined as those who were in stable condition at least 3 months before inclusion in the study, had no significant change in treatment regimen and had not been admitted to hospital due to disease progression;
* Fertile men and women of childbearing age voluntarily agree to take effective contraceptive measures from signing the ICF to 180 days after receiving the trial vaccine; Pregnancy tests for women of childbearing age during the screening period were negative.

Exclusion Criteria:

* Fever (> 14 years of age, axillary temperature ≥37.3℃; ≤14 years old, axillary temperature ≥37.5℃);
* SARS-CoV-2 nucleic acid test was positive during the screening period;
* Previous history of allergy to any vaccine or drug, such as: allergy, urticaria, severe skin eczema, dyspnea, laryngeal edema, angioneurotic edema, etc.;
* Those who have a history of immune deficiency diseases, major organ diseases, immune diseases [including Guillain-Barre syndrome (GBS), systemic lupus erythematosus, rheumatoid arthritis, asthenia or splenectomy caused by any circumstances, and other immune diseases that researchers believe may have an impact on the immune response], etc.;
* Currently suffering from severe or uncontrollable cardiovascular diseases, endocrine diseases, diseases of the blood and lymphatic systems, diseases of the liver and kidney, diseases of the respiratory system, diseases of the metabolic and skeletal systems or malignancies (other than basal cell carcinoma of the skin and carcinoma in situ of the cervix), such as severe heart failure, severe pulmonary heart disease, unstable angina, liver failure or uremia;
* The subjects are in an acute state of disease, such as acute onset of chronic heart failure, acute sore throat, hypertensive encephalopathy, acute pneumonia, acute renal insufficiency, acute cholecystitis, etc.;
* Anti-tuberculosis therapy is being used;
* Influenza vaccine within 14 days prior to vaccination or another type of vaccine within 28 days prior to vaccination;
* Use of immunosuppressant or immunomodulatory drugs for ≥14 days in the 6 months before enrollment, but short-term use of oral, inhaled and topical steroid hormones (≤14 days) is allowed;
* are pregnant or breastfeeding or plan to become pregnant during the study period;
* HIV-positive patients;

Ages: 3 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Safety endpoint: Incidence and severity of Solicited Adverse Events | Day 0~Day 7
  The incidence and severity of solicited adverse events on days 0-7 after inoculation with SCTV01E;
Immunogenicity endpoint 1: IgG total antibody concentration (ELISA) | Day 28
  IgG total antibody (ELISA) concentrations against SARS-CoV-2 prototype strains at 28 days post-vaccination and serum response rates (Geometric mean concentration [GMC], VOC/VOI based on epidemic variations can be tested);
Immunogenicity endpoint 2: Neutralizing antibody titer against SARS-CoV-2 Omicron variants (live virus neutralization test) | Day 28
  Geometric mean titer (GMT) and serum response rates at 28 days post-vaccination for neutralizing antibodies against SARS-CoV-2 Omicron variants (live virus neutralization test). VOC/VOI based on epidemic variations can be tested;

SECONDARY OUTCOMES:
Safety endpoint 1: Incidence and severity of Unsolicited Adverse Events | Day 0~Day 28
  Incidence and severity of unsolicited adverse events on days 0-28 after inoculation with SCTV01E;
Safety endpoint 2: Incidence and severity of Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) | Day 0~Day 180
  Incidence and severity of serious adverse events (SAEs) and adverse events of special interest (AESIs) within 180 days of vaccination with SCTV01E.
Immunogenicity endpoint 1: IgG total antibody concentration (ELISA) | Day 0~Day 180
  GMC and serum response rates of total IgG antibody (ELISA) against the prototype strain of SARS-CoV-2 on days 7, 14, 90 and 180 after inoculation with SCTV01E (other VOC/VOI can be increased depending on the epidemic situation);
Immunogenicity endpoint 2: Neutralizing antibody titer against SARS-CoV-2 Omicron variants (live virus neutralization test) | Day 0~Day 180
  GMT and serum response rates for neutralizing antibodies against SARS-CoV-2 Omicron variant (live virus neutralization test) on days 7, 14, 90 and 180 after inoculation with SCTV01E (other VOC/VOI can be tested depending on the epidemic situation);
Immunogenicity endpoint 3: T cell Response | Day 0~Day 90
  Number of T cell subsets secreting IFN-γ (for Th1) and IL-4 (for Th2) on day 7 and day 90 after SCTV01E in subjects ≥18 years old.

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Fengcai, Principal Investigator — Jiangsu Center for Disease Control and Prevention
Locations (4):
- China (4):
  - Lianshui County Center for Disease Control and Prevention, Lianshui, Jiangsu
  - Jiangsu Center for Disease Control and Prevention, Nanjing, Jiangsu
  - Taizhou Vaccine Clinical Research Center, Taizhou, Jiangsu
  - Dazhu County Center for Disease Control and Prevention, Dazhou, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tuekprakhon A, Nutalai R, Dijokaite-Guraliuc A, Zhou D, Ginn HM, Selvaraj M, Liu C, Mentzer AJ, Supasa P, Duyvesteyn HME, Das R, Skelly D, Ritter TG, Amini A, Bibi S, Adele S, Johnson SA, Constantinides B, Webster H, Temperton N, Klenerman P, Barnes E, Dunachie SJ, Crook D, Pollard AJ, Lambe T, Goulder P, Paterson NG, Williams MA, Hall DR; OPTIC Consortium; ISARIC4C Consortium; Fry EE, Huo J, Mongkolsapaya J, Ren J, Stuart DI, Screaton GR. Antibody escape of SARS-CoV-2 Omicron BA.4 and BA.5 from vaccine and BA.1 serum. Cell. 2022 Jul 7;185(14):2422-2433.e13. doi: 10.1016/j.cell.2022.06.005. Epub 2022 Jun 9. PMID 35772405
- [Background] WHO Coronavirus (COVID-19) Dashboard [EB/OL]. [2022-10-21]. https://covid19.who.int.
- [Background] COVID-19 vaccine tracker and landscape [EB/OL]. [2022-10-21]. https://www.who.int/publications/m/item/draft-landscape-of-covid-19-candidate-vaccines.
- [Background] WHO-COVID19 Vaccine Tracker [EB/OL]. [2022-10-21]. https://covid19.trackvaccines.org/agency/who/.
- [Background] 健康界. 中国疾控中心：新冠疫苗"加强针"仍免费接种；国务院联防联控机制：力争年底前完成3至11岁人群新冠疫苗接种|疫苗|接种|新闻|表示|人群|-健康界[EB/OL]. [2022-10-21]. https://www.cn-healthcare.com/articlewm/20211031/content-1279647.html.
- [Background] FDA. Coronavirus (COVID-19) Update: FDA Authorizes Moderna and Pfizer-BioNTech COVID-19 Vaccines for Children Down to 6 Months of Age [EB/OL]. [2022-10-21]. https://www.fda.gov/news-events/press-announcements/coronavirus-covid-19-update-fda-authorizes-moderna-and-pfizer-biontech-covid-19-vaccines-children.
- [Background] EverdayHEALTH-NEWS. BA.4 and BA.5 Omicron Subvariants Are Now Dominant in the U.S.[EB/OL]. [2022-10-21]. https://www.everydayhealth.com/coronavirus/ba4-and-ba5-have-become-dominant-omicron-subvariants-in-the-us/.